CLINICAL TRIAL: NCT06150027
Title: A Randomized Comparative Prospective Multicenter Study of the Efficacy of a Systematic Referral to Palliative Care of Patients Who Need for Palliative Care During an Unscheduled Visit in Comprehensive Anticancer Centers
Brief Title: Efficacy of a Systematic Referral to Palliative Care of Patients Who Need for Palliative Care During an Unscheduled Visit in Comprehensive Anticancer Centers
Acronym: PALLU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ET22-175
Record Dates: First submitted 2023-11-17; First posted 2023-11-29 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Cancer; Emergencies
Keywords: Early palliative care; Cancer; Aggressiveness of care; Emergency
MeSH Terms: conditions — Neoplasms; Emergencies

STUDY DESIGN:
Intervention Model Description: Randomization (ratio 1:1) will be stratified according to the investigation center and pre-existing follow-up by pain management team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard (No Intervention): Conventional strategy: patients will be managed regardless of their PALLIA-10 score. The need for additional care, including palliative care, will be assessed by the team in charge of the patient, as per routine practice.
- Experimental (Experimental): Experimental strategy: patients will be systematically referred to a palliative care team.
  Interventions: Other: Systematic referral to a palliative care team

INTERVENTIONS:
Other: Systematic referral to a palliative care team — Patients randomized in the experimental arm will be systematically referred to a palliative care team.
  A follow-up in palliative care will be initiated for all within a maximum of 15 days after the date of randomization.
  Arms: Experimental

SUMMARY:
This is a randomized, multicenter, prospective, phase III study conducted in daily emergency rooms of French Regional Comprehensive Cancer Centers.

In the standard arm, patients will be managed regardless of their PALLIA-10 score, following conventional strategy. In the experimental arm, patients will be systematically referred to a palliative care team.

DETAILED DESCRIPTION:
This is a randomized, multicenter, prospective, phase III study conducted in daily emergency rooms of French Regional Comprehensive Cancer Centers.

All patients undergoing a visit in the daily emergency room of a participating center and who need for palliative management (PALLIA 10 score > 3/10) will be considered for inclusion in the PALLU study. After signing the written informed consent, patients will be randomized (1:1 ratio) in one of the following arms:

* Standard arm : conventional strategy; patients will be managed regardless of their PALLIA-10 score. The need for additional care, including palliative care, will be assessed by the team in charge of the patient, as per routine practice.
* Experimental arm : experimental strategy; patients will be systematically referred to a palliative care team.

Randomization will be stratified according to the investigation center and pre-existing follow-up by pain management team.

The difference of intervention will lie in the fact that patients will be referred or not to a palliative care team but patients from the standard arm may receive palliative care as deemed necessary by the medical oncology team. In this case, the content of palliative care for patients included in both groups will be identical.

The end of the study will be the Last Patient Last Visit (LPLV), defined as the date of the 12-month visit of the last patient still alive or when the 192nd death has occurred, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years at the day of consenting to the study;
* Confirmed diagnosis of any type of solid or haematology tumours, with or without Current oncological treatment, such as chemotherapy, immunotherapy, targeted therapy, etc;
* Unscheduled admission in a French Regional Comprehensive Anti-Cancer Centre due to an acute, unpredictable, intercurrent event related to cancer, its therapies or a comorbidity;
* Patient for whom disease is considered as not curable;
* PALLIA-10 Score > 3/10;
* Willingness and ability to comply with the study requirements;
* Signed and dated informed consent indicating that the patient has been informed of all the aspects of the trial prior to enrolment;
* Patient must be covered by a medical insurance.

Exclusion Criteria:

* Patient without consciousness, unable to provide a written informed consent (context of emergency);
* Patient treated with a curative intent;
* Previous randomization in this clinical study;
* Patients already followed-up by a palliative care team;
* Life expectancy shorter than 1 month, as per the emergency units' staff judgement.
* Any medical or psychosocial condition that would compromise the patient's compliance to the study visits or would likely interfere with the completion of Patient-Reported Outcomes.
* Patients under tutorship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Aggressiveness of care near the end of life | From date of randomization until the date of death from any cause, assessed up to 30 months
  Percentage and number of patients who meet at least one of the following criteria :
  * More than 1 hospitalization in the last 30 days of life;
  * More than 1 visit in an emergency unit in the last 30 days of life;
  * More than 14 days in hospital in the last 30 days of life;
  * Hospitalization in a resuscitation unit in the last 30 days of life;
  * Treatment with systemic anticancer therapy in the last 14 days of life;
  * New systemic anticancer therapy regimen starting in the last 30 days of life;
  * Patients dying in an acute care setting.

SECONDARY OUTCOMES:
More than 1 hospitalization in the last 30 days of life | From date of randomization until the date of death from any cause, assessed up to 48 months
  Percentage and number of patients having more than 1 hospitalization in the last 30 days of life
More than 1 visit in an emergency unit in the last 30 days of life | From date of randomization until the date of death from any cause, assessed up to 30 months
  Percentage and number of patients having more than 1 visit in an emergency unit in the last 30 days of life
More than 14 days in hospital in the last 30 days of life | From date of randomization until the date of death from any cause, assessed up to 30 months
  Percentage and number of patients having more than 14 days in hospital in the last 30 days of life
Hospitalization in a resuscitation unit in the last 30 days of life | From date of randomization until the date of death from any cause, assessed up to 30 months
  Percentage and number of patients having a hospitalization in a resuscitation unit in the last 30 days of life
Treatment with chemotherapy in the last 14 days of life | From date of randomization until the date of death from any cause, assessed up to 30 months
  Percentage and number of patients having a treatment with chemotherapy in the last 14 days of life
New chemotherapy regimen starting in the last 30 days of life | From date of randomization until the date of death from any cause, assessed up to 30 months
  Percentage and number of patients having a new chemotherapy regimen starting in the last 30 days of life
Death in an acute care setting | At the date of death from any cause, assessed up to 30 months
  Percentage and number of patients dying in an acute care setting
Medical resources mobilized in terms of palliative care | From date of randomization until the date of death from any cause, assessed up to 30 months
  Medical resources mobilized in terms of palliative care (psychologist, social worker, nutritional counselling, etc.) will be described for the interventional group in terms of number and percentage of patients with at least one consultation with each specialist
Health-related quality of life using the FACT-G7 cancer specific questionnaire | At inclusion, 3 months, 6 months, 9 months and at 12 months
  The total score ranges from 0 and 28, with a higher score indicates better quality of life. Scores will be described per randomized group at each measurement time (inclusion,3 months and 6 months) using same criteria as for other quantitative variables (number of observations, mean, standard deviation, median, minimum and maximum values).
Health-related quality of life using the HADS | At inclusion, 3 months, 6 months, 9 months and at 12 months
  One score is generated for anxiety and one score for depression on a 0 to 21 points, with a higher score indicates higher level of trouble. Scores will be described per randomized group at each measurement time (inclusion,3 months and 6 months) using same criteria as for other quantitative variables (number of observations, mean, standard deviation, median, minimum and maximum values). Number and percentage of patients without anxiety or depression trouble (i.e. with a score of 7 or lower), moderate trouble (score between 8 to 10) and severe trouble (score of 11 or more) will be reported.
Symptoms of cancer disease using the Edmonton Symptoms Assessment System (ESAS) symptom scores | From date of randomization until the date of death from any cause, assessed up to 30 months
  Pain, tiredness, drowsiness, nausea, lack of appetite, depression, anxiety, shortness of breath, and wellbeing and patient-specific symptoms are each described on a scale ranging from 0 to 10 (10 being the worst). The mean change in symptoms will be estimated from baseline and at each follow-up time. The ESAS symptom scores will be calculated according to the authors' recommendations and described per randomized group at each time point by mean, standard deviation, median and range.
Place of death | At the date of death from any cause, assessed up to 30 months
  Hospital and type of unit or home will be described per randomized group
Overall Survival | At the date of death from any cause, assessed up to 30 months
  Defined as the time from the date of inclusion to the date of death due to any cause.

OTHER OUTCOMES:
Health improvement (Life Year gained) | 12 months from randomization
  Health improvement will be measured in Life Year (LY) gained.
Health improvement (Quality-Adjusted Life Years gained) | 12 months from randomization
  Health improvement will be measured in Quality-Adjusted Life Years (QALY) gained, based on the EQ-5D-5L assessments, performed at inclusion, 3 months, 6 months, 9 months and at 12 months. For EQ-5D-5L, 5 attributes will therefore be investigated: mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. Each attributes having five levels. The score falls on the 0.0 (dead) to 1.0 (perfect health) value scale.
  The value set for the EQ-5D-5L based on societal preferences of the French population will be used. QALYs will be calculated as the sum of QALY of each of the periods weighted by it respective probability. Effects will be also not discounted.
Mean Total Costs | 12 months from randomization
  Mean total costs associated with each strategy, including hospital care, outpatient care, medical goods, transport, and palliative support.
Impact of clinical variables on cost | 12 months from randomization
  Multiple regression analyses will be performed to examine the correlation between costs and a range of potentially explanatory clinical variables
Impact of patient variables on cost | 12 months from randomization
  Multiple regression analyses will be performed to examine the correlation between costs and a range of potentially explanatory patient variables
Sensitivity Analyses | 12 months from randomization
  One-way sensitivity analyses varying all cost items by minimal and maximal values observed in the sample
Incremental Cost-Effectiveness Ratio (ICER) per QALY gained | 12 months from randomization
  The ICER will compare the cost per QALY gained between the experimental strategy and the conventional strategy.
  QALY gained will be based on the EQ-5D-5L assessments, performed at inclusion, 3 months, 6 months, 9 months and at 12 months. For EQ-5D-5L, 5 attributes will therefore be investigated: mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. Each attributes having five levels. The score falls on the 0.0 (dead) to 1.0 (perfect health) value scale.
  The value set for the EQ-5D-5L based on societal preferences of the French population will be used. QALYs will be calculated as the sum of QALY of each of the periods weighted by it respective probability. Effects will be also not discounted.
Incremental Cost-Effectiveness Ratio (ICER) per LY gained | 12 months from randomization
  The ICER will compare the cost per LY gained between the experimental strategy and the conventional strategy.
Emergency healthcare professionals' perceptions of early palliative care before the beginning of recruitment | Before the beginning of recruitmentof in their centre
  Described by the potential factors limiting or facilitating the referral of patients to palliative caregivers. Descriptive analyses will be done. Quantitative variables will be described with mean (standard deviation) and median (min-max). Qualitative variables will be described with numbers and percentages.

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle CHVETZOFF, MD,PhD, Principal Investigator — Centre Leon Berard
Locations (6):
- France (6):
  - Centre Léon Bérard, Lyon
  - ICM Val d'Aurelle, Montpellier
  - Institut Curie - Paris, Paris
  - Institut Curie - Saint Cloud, Saint-Cloud
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
In the patient information sheet and informed consent form, the participants do not agree to share their individual personal data.

REFERENCES:
- [Derived] Chvetzoff G, Anota A, Perrier L, Gautier J, Bouleuc C, Moreau P, Thomaso M, Le Divenah G, Henry A, Francois M, Massiani MA, Mateus C, Merad M, Bissuel L, Baudry AS, Christophe V, Russias B, Perol D. Systematic referral to palliative care in patients attending dedicated emergency units from French comprehensive anticancer centres: the prospective multicentre randomised comparative clinical trial PALLU. BMJ Open. 2025 Aug 24;15(8):e101299. doi: 10.1136/bmjopen-2025-101299. PMID 40850913